CLINICAL TRIAL: NCT04380285
Title: Treating Heel Pain Associated With Plantar Fasciitis in Adults: A Randomized Clinical Trial of Hard Versus Modified Soft Custom Orthotics and Heel Pads
Brief Title: Treating Heel Pain in Adults: A Randomized Clinical Trial of Hard Versus Soft Orthotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deborah Seligman, MSc., B.Sc.O.T. (Other)
Responsible Party: Sponsor-Investigator, Deborah Seligman, MSc., B.Sc.O.T., Occupational Therapist, University of Toronto
Organization: University of Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #9964
Record Dates: First submitted 2020-04-28; First posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Heel Pain Syndrome
Keywords: Foot; Heel Pain; Plantar Fasciitis; Orthotic Devices
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Intervention Model Description: The study design was a randomized clinical trial.The study was completed when the target number of recruitments was reached. Prior to randomization to treatment groups, patients were stratified by age (younger adults: 18 - 64 years and older adults: 65 years and older) in blocks of four to ensure that there were an equal number of participants receiving soft versus hard orthotics in each age group.
Who Masked: Outcomes Assessor
Masking Description: The research assistant was blinded to the type of orthotic provided to the participant to prevent possible bias during administration of the post treatment questionnaire.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1. Custom heel pads and modified soft molded orthotics (Active Comparator): Modified soft custom orthotics supported in the medial longitudinal arches and medial shock absorbing heel pads with customized cutout at the point corresponding to the heel pain
  Interventions: Device: Custom heel pads and modified soft molded orthotics
- Group 2. Custom hard orthotics (Active Comparator): Custom hard orthotics made from a positive mold of a foot in neutral position, with arch support and medial heel postings.
  Interventions: Device: Custom hard orthotic

INTERVENTIONS:
Device: Custom heel pads and modified soft molded orthotics
  Arms: Group 1. Custom heel pads and modified soft molded orthotics
Device: Custom hard orthotic
  Arms: Group 2. Custom hard orthotics

SUMMARY:
Objectives: This study compared the effectiveness of soft versus hard orthotics in treating heel pain and plantar fasciitis in adults. It also compared the level of function after orthotic use, cost and number of visits for orthotics and explored if age was a factor in orthotic effectiveness.

DETAILED DESCRIPTION:
Design: This randomized clinical trial included 44 adults (18+) with heel pain and plantar fasciitis. Participants received hard or soft customized orthotics and rated their pain intensity, pain interference and function, pre and post orthotic use. Scores were analyzed with repeated measures ANOVA. Analysis of age used repeated measures ANOVA. Costs were compared using t-test and number of visits was compared using Wilcoxon Rank Sum.

ELIGIBILITY:
Inclusion Criteria:

* sample of convenience from the hospital and private clinic. The participants had heel pain associated with plantar fasciitis. Participants could describe and report changes in their pain

Exclusion Criteria:

* Those excluded were non-ambulatory (unable to walk greater than 25 meters) orchid spasticity due to a neurological disorder. Others excluded were non-communicative, had cognitive impairment or were unable to complete a questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2003-01 (Actual); Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory: a sub-scale from this measurement tool measuring pain intensity. Change in pain intensity is being assessed using this measurement tool pre and post treatment. | This questionnaire was administered on the initial visit and then 6 weeks after orthotics were provided.
  Measures pain intensity on a numeric rating scale with anchors of 'no pain' (0) to 'pain as bad as you can imagine' (10)

SECONDARY OUTCOMES:
Brief Pain Inventory: a sub-scale from this measurement tool measuring pain interference with activity and level of function. Change in pain interference is being assessed using this measurement tool pre and post treatment. | This questionnaire was administered on the initial visit and then 6 weeks after orthotics were provided.
  Pain interference was rated on the following items: general activity, walking, work, relations with other people, mood, sleep and enjoyment of life, using a numeric scale with anchors 'does not interfere (0) to 'completely interferes' (10)
Late Life Function and Disability Instrument (Late Life FDI): Function component. Change in function is being assessed using this measurement tool pre and post treatment. | This questionnaire was administered on the initial visit and then 6 weeks after orthotics were provided.
  It rates one's ability to do a wide variety of activities that involve basic upper and lower extremity function, such as reaching, standing and bending as well as higher levels of physical endurance such as walking and climbing stairs.It is a 32 item self-report questionnaire with five response categories and a score ranging from 32 to 160.

CONTACTS AND LOCATIONS:
Overall Officials: Aileen Davis, PhD,BScPT, Principal Investigator — University of Toronto

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, measurement tools, interventions used.
Supporting Information: Study Protocol
Time Frame: 6 months after publication for a period of 6 months
Access Criteria: can email principle investigator/author directly

REFERENCES:
- [Derived] Seligman DAR, Dawson D, Streiner DL, Seligman DJ, Davis A. Treating Heel Pain in Adults: A Randomized Controlled Trial of Hard vs Modified Soft Custom Orthotics and Heel Pads. Arch Phys Med Rehabil. 2021 Mar;102(3):363-370. doi: 10.1016/j.apmr.2020.10.124. Epub 2020 Nov 18. PMID 33217374